CLINICAL TRIAL: NCT03010254
Title: A Prospective, Randomized, Controlled, Multi-Center Clinical Study of the ACRYSOF® IQ Extended Depth of Focus (EDF) IOL
Brief Title: A Clinical Study of the ACRYSOF® IQ EDF Intraocular Lens (IOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILI875-C001
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- DFT015 (Experimental): ACRYSOF® IQ Extended Depth of Focus Intraocular lens (IOL), bilateral implantation
  Interventions: Device: ACRYSOF® IQ Extended Depth of Focus IOL; Procedure: Cataract surgery
- SN60WF (Active Comparator): ACRYSOF® IQ Monofocal IOL, bilateral implantation
  Interventions: Device: ACRYSOF® IQ Monofocal IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: ACRYSOF® IQ Extended Depth of Focus IOL — Implantable IOL intending to extend the depth of focus and provide continuous functional vision from distance to near while maintaining distance vision and a visual disturbance profile comparable to a monofocal IOL; intended for long-term use over the lifetime of the pseudophakic subject
  Other Names: Model DFT015
  Arms: DFT015
Device: ACRYSOF® IQ Monofocal IOL — Monofocal IOL implanted for long-term use over the lifetime of the pseudophakic subject
  Other Names: Model SN60WF
  Arms: SN60WF
Procedure: Cataract surgery — IOL bilateral implantation

SUMMARY:
The purpose of the study is to demonstrate the safety and performance of the ACRYSOF® IQ EDF IOL.

DETAILED DESCRIPTION:
Both eyes will be implanted. The second eye implantation will occur a minimum of 7 calendar days and a maximum of 28 calendar days from the first eye implantation.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an Independent Ethics Committee (IEC)/ Institutional Review Board (IRB) approved Informed Consent Form;
* Diagnosed with cataract in both eyes;
* Planned cataract removal by routine small incision surgery;
* Calculated IOL power is within the clinical study supply range (18.0-25.0 diopter (D) in 0.5 D steps);
* Preoperative regular astigmatism of less than 1.0 D.

Exclusion Criteria:

* Pregnancy or lactation current or planned during the course of the study;
* History of anterior segment (corneal, anterior chamber, sulcus) or posterior segment (uveal, vitreo-retinal) pathology including retinal vascular occlusive disease, retinal detachment or peripheral retinal laser photocoagulation, age-related macular degeneration (ARMD), glaucoma (uncontrolled or controlled with medication) or ocular hypertension, diabetic retinopathy, retinitis pigmentosa and any optic nerve pathology.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Clinical Manager, GCRA, Study Director — Alcon Research
Locations (18):
- Australia (4):
  - Alcon Investigative Site, Sydney, New South Wales
  - Alcon Investigative Site, Southport, Queensland
  - Alcon Investigative Site, Footscray, Victoria
  - Alcon Investigative Site, Hawthorn East, Victoria
- Canada (5):
  - Alcon Investigative Site, Vancouver, British Columbia
  - Alcon Investigative Site, Mississauga, Ontario
  - Alcon Investigative Site, Toronto, Ontario
  - Alcon Investigative Site, Boisbriand, QU
  - Alcon Investigative Site, Québec, QU
- Spain (5):
  - Alcon Investigative Site, Sant Cugat del Vallès, BCN
  - Alcon Investigative Site, Jerez de la Frontera, Cadiz
  - Alcon Investigative Site, Barcelona
  - Alcon Investigative Site, Madrid
  - Alcon Investigative Site, Valencia
- United Kingdom (4):
  - Alcon Investigative Site, Dartford, Kent
  - Alcon Investigative Site, Essex
  - Alcon Investigative Site, London
  - Alcon Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bala C, Poyales F, Guarro M, Mesa RR, Mearza A, Varma DK, Jasti S, Lemp-Hull J. Multicountry clinical outcomes of a new nondiffractive presbyopia-correcting IOL. J Cataract Refract Surg. 2022 Feb 1;48(2):136-143. doi: 10.1097/j.jcrs.0000000000000712. PMID 34288635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 21 investigative sites located in Australia, Canada, Spain and the United Kingdom.
Pre-assignment Details: A total of 322 subjects were enrolled in the study, out of which 39 subjects exited due to screen failure and 1 subject discontinued due to site being closed before actual screening visit and randomization. This reporting group includes all randomized subjects.
Period: Overall Study
Arm/Group | DFT015 | SN60WF
Started (All randomized subjects) | 159 | 123
Attempted Implantation | 156 | 120
Successful Implantation | 156 | 120
Completed | 152 | 118
Not Completed | 7 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Population: This analysis population included all randomized eyes with successful IOL implantation (All-Implanted Analysis Set).
Groups:
- DFT015: ACRYSOF® IQ Extended Depth of Focus IOL, bilateral implantation
- Total: Total of all reporting groups
Arm/Group | DFT015 | SN60WF | Total
Number analyzed (Participants) | 156 | 120 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (7.37) | 69.7 (7.54) | 69.7 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 65 | 159
  Male | 62 | 55 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 25 | 56
  Not Hispanic or Latino | 107 | 79 | 186
  Unknown or Not Reported | 18 | 16 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 8 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 129 | 101 | 230
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Monocular Photopic Distance Corrected Intermediate Visual Acuity (DCIVA) at 66 Centimeters (cm)
Description: Visual Acuity (VA) was assessed monocularly (each eye separately) under photopic (well-lit) conditions using best distance correction (distance refraction) and high contrast, Early Treatment Diabetic Retinopathy Study (ETDRS) chart at 66 cm from spectacle plane. It was measured in logarithm of the minimum angle of resolution (logMAR), with 0.02 logMAR increment corresponding to a single letter or 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. This analysis was prespecified for the first operative eye.
Time Frame: Month 3 (70-100 days post second eye implantation)
Population: All-Implanted Analysis Set
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 153 | 115
Number analyzed (Eyes) | 153 | 115
logMAR | 0.175 (0.0137) | 0.313 (0.0158)
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Test type: Superiority; p < 0.001, t-test, 2 sided — 2-sided p-value reported. A hypothesis test was based on a two sample t-test, with a type I error rate of 0.025, 1-sided; Least Squares Mean Difference = -0.138, 95% CI 2-sided [-0.180 to -0.097], Standard Error of Mean 0.0210 — Least squares mean difference (DFT015 - SN60WF)

2. Primary Outcome: Percentage of Subjects With Ocular Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device (test article). Ocular AEs are events localized to the eye. Cumulative and persistent serious adverse events as defined by ISO 11979-7:2014 were collected for Model DFT015 first and second eyes. No formal statistical hypothesis testing was planned.
Time Frame: Day 0 (first operative eye visit) up to Month 6 (120-180 days post second eye implantation)
Population: This analysis population included all eyes with attempted IOL implantation (successful or aborted after contact with the eye) (Safety Analysis Set). This outcome measure was pre-specified for the ACRYSOF® IQ Extended Depth of Focus IOL DTF015 only.
Measure: Number; unit: percentage of subjects
Units Other Than Participants: Eyes
Groups:
- DFT015 First Eye: All eyes with attempted test article implantation (successful or aborted after contact with the eye) in the first implanted eye
- DFT015 Second Eye: All eyes with attempted test article implantation (successful or aborted after contact with the eye) in the second implanted eye
Arm/Group | DFT015 First Eye | DFT015 Second Eye
Number analyzed (Participants) | 156 | 154
Number analyzed (Eyes) | 156 | 154
percentage of subjects
  Cumulative: Cystoid macular oedema | 0.6 | 0.0
  Cumulative: Hypopyon | 0.0 | 0.0
  Cumulative: Endophthalmitis | 0.0 | 0.0
  Cumulative: Lens dislocated from posterior chamber | 0.0 | 0.0
  Cumulative: Pupillary block | 0.0 | 0.0
  Cumulative: Retinal detachment | 0.0 | 0.0
  Cumulative: Secondary surgical intervention | 0.6 | 0.6
  Persistent: Corneal stroma oedema | 0.0 | 0.0
  Persistent: Cystoid macular oedema | 0.0 | 0.0
  Persistent: Iritis | 0.0 | 0.0
  Persistent: Raised IOP requiring treatment | 0.0 | 0.0

3. Secondary Outcome: Monocular Photopic Best Corrected Distance Visual Acuity (BCDVA) at 4 Meters (m)
Description: VA was tested monocularly under photopic conditions using the correction obtained from the manual manifest refraction and 100% contrast, ETDRS charts at a distance of 4 m from the spectacle plane. VA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter or 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. This analysis was prespecified for the first operative eye.
Time Frame: Month 3 (70-100 days post second eye implantation)
Population: All-Implanted Analysis Set
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 153 | 115
Number analyzed (Eyes) | 153 | 115
logMAR | -0.007 (0.0076) | -0.044 (0.0087)
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Test type: Non-Inferiority — Non-inferiority margin was 0.1 logMAR; Least Squares Mean Difference = 0.037, 97.5% CI 1-sided [upper limit 0.059], Standard Error of Mean 0.0115 — Least squares mean difference (DFT015 - SN60WF).The 1-sided 97.5% Upper Confidence Limit is presented

4. Secondary Outcome: Monocular Photopic Distance Corrected Near Visual Acuity (DCNVA) at 40 cm
Description: VA was tested monocularly under photopic conditions using best distance correction (distance refraction) and high contrast, ETDRS chart set at 40 cm from the spectacle plane using the near point rod. VA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter or 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. This analysis was prespecified for the first operative eye.
Time Frame: Month 3 (70-100 days post second eye implantation)
Population: All-Implanted Analysis Set
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 153 | 115
Number analyzed (Eyes) | 153 | 115
logMAR | 0.420 (0.0142) | 0.510 (0.0163)
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Test type: Superiority; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.090, 95% CI 2-sided [-0.133 to -0.048], Standard Error of Mean 0.0216 — Least squares mean difference (DFT015 - SN60WF)

5. Secondary Outcome: Monocular Photopic Distance Corrected Depth of Focus Assessed by the Mean Defocus Curve
Description: Depth of focus was assessed at 4 meters under photopic (well-lit) conditions using best corrected distance refraction, added defocus and 100% contrast ETDRS charts. VA was measured between +1.50 Diopter (D) and -2.50 D in 0.5 D defocus steps, except in the region from +0.50 D through -0.50 D, which was assessed in 0.25 D steps. VA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter or 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. The depth of focus was estimated as the dioptric range between zero defocus and the first point on the negative lens induced mean defocus curve that crosses the 0.2 logMAR using a linear interpolation. A lower numeric value represents better VA. This analysis was pre-specified for the first operative eye. No formal statistical hypothesis testing was planned.
Time Frame: Month 3 (70-100 days post second eye implantation)
Population: This analysis population included all eyes successfully implanted that had at least 1 postoperative visit, no macular degeneration at any time, and no major protocol violations (Best-case Analysis Set). Number analyzed is the number of subjects/eyes with data available for analysis at specified defocus.
Measure: Number; unit: diopter
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 151 | 104
Number analyzed (Eyes) | 151 | 104
diopter | 1.61 | 1.09
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Test type: Other; Hypothesis testing was not pre-specified; Mean difference in depth of focus = 0.52 — Mean difference in depth of focus (DFT015 - SN60WF)

6. Secondary Outcome: Monocular Mesopic Contrast Sensitivity at 12 Cycles Per Degree (Cpd)
Description: Contrast sensitivity (i.e., the ability to detect objects by distinguishing them from their background) was assessed monocularly with the subject's best spectacle correction under mesopic (low, but not quite dark) conditions at a distance of 8 feet (2.45 m) from the eye at a spatial frequency of 12 cpd using the Vector Vision CSV 1000-HGT with and without a glare source. Raw scores from contrast sensitivity testing were transformed to log units. A higher numeric value represented better contrast sensitivity. This analysis was prespecified for the first operative eye.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: All-Implanted Analysis Set. Number analyzed is the number of subjects/eyes with data available for analysis at without glare and with glare assessments.
Measure: Least Squares Mean (Standard Error); unit: log unit
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 156 | 120
Number analyzed (Eyes) | 156 | 120
log unit
  Without Glare: number analyzed (Participants) | 152 | 118
  Without Glare: number analyzed (Eyes) | 152 | 118
  Without Glare | 0.799 (0.0364) | 0.978 (0.0413)
  With Glare: number analyzed (Participants) | 152 | 118
  With Glare: number analyzed (Eyes) | 152 | 118
  With Glare | 0.794 (0.0357) | 0.975 (0.0406)
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Without glare; Test type: Non-Inferiority — Non-inferiority margin was -0.15 log unit; Least Squares Mean Difference = -0.179, 97.5% CI 1-sided [lower limit -0.287], Standard Error of Mean 0.0551 — Least squares mean difference (DFT015 - SN60WF). The 1-sided 97.5 Lower Limit Confidence Interval is presented
Statistical Analysis 2: Comparison: DFT015 vs SN60WF; With glare; Test type: Non-Inferiority — Non-inferiority margin was -0.15 log unit; Least Squares Mean Difference = -0.181, 97.5% CI 1-sided [lower limit -0.287], Standard Error of Mean 0.0541 — Least squares mean difference (DFT015 - SN60WF). The 1-sided 97.5 Lower Limit Confidence Interval is presented

7. Secondary Outcome: Percentage of Subjects Who Respond "Never" to Question 1 of the Spectacle Use Questionnaire: "How Often Do You Wear Eyeglasses for Any Purpose?"
Description: Proportion of subjects was reported as a percentage. No formal statistical hypothesis testing was planned.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: All-Implanted Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 106 | 80
percentage of subjects | 30.2 | 10.0
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Test type: Superiority; Difference in percentage = 20.2, 95% CI 2-sided [8.77 to 31.04] — 95% CI for the difference (DFT015 - SN60WF) is estimated using Miettinen-Nurminen method (1985)

8. Secondary Outcome: Percentage of Subjects Who Respond "Never" to Question 3 of the Spectacle Use Questionnaire: "How Often Do You Wear Eyeglasses for Intermediate Tasks (e.g., Computer)?"
Description: No formal statistical hypothesis testing was planned.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: All-Implanted Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 106 | 80
percentage of subjects | 75.5 | 53.8
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Test type: Superiority; Percent difference = 21.7, 95% CI 2-sided [7.92 to 35.06] — 95% CI for the difference (DFT015 - SN60WF) is estimated using Miettinen-Nurminen method (1985)

ADVERSE EVENTS:
Time Frame: Pre-operation (Day -28) up to Day 120-180 (post second eye implantation), up to 8 months
Description: An AE was any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. Safety Analysis Set. "At Risk" population of preoperative and systemic AEs is reported in units of subjects; all other AE populations are reported in units of eyes.
Groups:
- Preoperative: All subjects in the safety analysis set prior to initiation of treatment
- DFT015 Systemic: All subjects with attempted test article implantation (successful or aborted after contact with the eye)
- SN60WF First Eye: All eyes with attempted control article implantation (successful or aborted after contact with the eye) in the first implanted eye
- SN60WF Second Eye: All eyes with attempted control article implantation (successful or aborted after contact with the eye) in the second implanted eye
- SN60WF Systemic: All subjects with attempted control article implantation (successful or aborted after contact with the eye)
Arm/Group | Preoperative | DFT015 First Eye | DFT015 Second Eye | DFT015 Systemic | SN60WF First Eye | SN60WF Second Eye | SN60WF Systemic
All-Cause Mortality (participants affected / at risk) | 0/276 | 0/156 | 0/154 | 0/156 | 0/120 | 0/119 | 0/120
Serious Adverse Events (participants affected / at risk) | 1/276 | 2/156 | 2/154 | 3/156 | 2/120 | 0/119 | 9/120
Other Adverse Events (participants affected / at risk) | 0/276 | 0/156 | 0/154 | 0/156 | 0/120 | 0/119 | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative (N=276) | DFT015 First Eye (N=156) | DFT015 Second Eye (N=154) | DFT015 Systemic (N=156) | SN60WF First Eye (N=120) | SN60WF Second Eye (N=119) | SN60WF Systemic (N=120)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystoid macular oedema (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Posterior capsule rupture (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Refraction disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitreous loss (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intraocular lens repositioning (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Keratomileusis (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitrectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT03010254/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT03010254/SAP_001.pdf